CLINICAL TRIAL: NCT02350166
Title: Short-term Effects of Laparoscopic-assisted Small-incision Surgery Versus Conventional Laparotomy in Treatment of Resectable Colorectal Liver Metastasis
Brief Title: Short-term Effects of LASI Surgery Versus Conventional Laparotomy for Colorectal Liver Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor of the West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sLRC-201312
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; hepatectomy; laparoscopic surgery; laparotomy; complications
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic group (Experimental): Laparoscopic group, laparoscopic surgery or laparoscopic-assisted small-incision for resection of laparoscopic colorectal tumor combined with synchronously small-incision open resection of liver metastasis
  Interventions: Procedure: laparoscopic surgery
- Conventional group (No Intervention): Conventional group, conventional laparotomy for simultaneously resection of both primary colorectal tumor and liver metastasis

INTERVENTIONS:
Procedure: laparoscopic surgery — laparoscopic-assisted small-incision surgery
  Arms: Laparoscopic group

SUMMARY:
Surgical resection is still recommended as the optional treatment for colorectal liver metastasis (CLM) patients. There are two main concerns for resectable colorectal liver metastasis which remain controversial: surgical time and surgical type. As for the former, synchronous resection of primary colorectal tumor and liver metastasis, with the reason of fare overall survival rate and absence of a second surgery, has gained wide population from gastrointestinal surgeons who believe it will bring benefits to CLM patients. With regard to surgical type, Open liver resection is the optimum choice for CLM patients no matter what the metastasis profile is. And for management of primary tumor, laparoscopic procedure is mature in surgical skill and has been evidenced equivalent overall survival rate compared with open resection. So, primary colorectal tumor resection could be either open or laparoscopic procedure. Therefore, the investigators team conducted the controlled trial to compare two surgical procedures in treatment of resectable colorectal liver metastasis. Patients will be randomly assigned into conventional laparotomy group for simultaneously resection of both primary colorectal tumor and liver metastasis, or laparoscopic-assisted small-incision group for resection of laparoscopic colorectal tumor combined with synchronously small-incision open resection of liver metastasis. The aim of this trial is to observing short-term operative effects after surgeries.

DETAILED DESCRIPTION:
Nowadays, colorectal liver metastasis (CLM) is gaining wide population from multi-disciplinary doctors including gastroenterologists, oncologists, and hepatic doctors for its increasing incidence and poor prognosis. Nearly, 15%-25% of colorectal cancer patients present with simultaneous liver metastasis at the time of diagnosis and 20%-35% patients are evaluated with primary tumor and liver metastasis resectable synchronously. Although the use of chemotherapy regimen has been certified favorable outcomes, surgical resection is still recommended as the optional treatment for CLM patients. However, there are two main concerns for resectable colorectal liver metastasis which remain controversial: surgical time and surgical type. As for the former, a latest evidence shows synchronous resection of primary colorectal tumor and liver metastasis, with the reason of fare overall survival rate and absence of a second surgery. Moreover, an increasing number of surgeons favor synchronous resection from their initial experience and they believe it will bring benefits to CLM patients.

With regard to surgical type, although laparoscopic liver resection has been proven feasible, safe and efficient in management of liver metastasis, this procedure is limited in selected patients such as tumor size less than 10 centimeters or located in left liver. In addition, laparoscopic liver resection is technically difficult which is applied in most medical centers. So open liver resection may be the optimum choice for CLM patients no matter what the metastasis profile is. In the management of primary tumor, laparoscopic procedure is mature in surgical skill and has been evidenced equivalent overall survival rate compared with open resection. A research conducted by Arezzo also confirms lower 30-day morbidity of laparoscopic colorectal cancer resection. Unlike liver metastasis resection, primary colorectal tumor resection could be either open or laparoscopic procedure.

Therefore, the investigators team conducted the controlled trial to compare two surgical procedures in treatment of resectable colorectal liver metastasis. Patients will be randomly assigned into conventional laparotomy group for simultaneously resection of both primary colorectal tumor and liver metastasis, or laparoscopic-assisted small-incision group for resection of laparoscopic colorectal tumor combined with synchronously small-incision open resection of liver metastasis. The aim of this trial is to observing short-term operative effects after surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed resectable upper rectal cancer, sigmoid cancer, and left colon cancer
2. MRI/CT confirmed resectable liver metastasis after muti-disciplinary team assessment
3. No evidence of other metastasis
4. Organs function well to tolerance simultaneous surgery, especially liver function
5. No special treatment before surgery
6. Informed consent was written

Exclusion Criteria:

1. Right colon cancer and transverse colon cancer
2. Pregnant or lactating women
3. A history of malignant tumor within 5 years
4. There was contraindication for operation
5. Discovery of metastasis in other organs in the operation
6. With mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
30-day complications | Postoperative 30 days
  Postoperative 30-day complications including anastomotic leakage, infection, and bile leakage

SECONDARY OUTCOMES:
Pain score | Postoperative 7 days
  Postoperative pain assessment
Hospital time | an expected average of 7 days
  Postoperative stay in hospital
C-reactive protein | Postoperative 5 days
  serum C-reactive protein level after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD,PhD, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - West China hospital, Sichuan University, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Siegel R, Ward E, Brawley O, Jemal A. Cancer statistics, 2011: the impact of eliminating socioeconomic and racial disparities on premature cancer deaths. CA Cancer J Clin. 2011 Jul-Aug;61(4):212-36. doi: 10.3322/caac.20121. Epub 2011 Jun 17. PMID 21685461
- [Background] Van Cutsem E, Nordlinger B, Adam R, Kohne CH, Pozzo C, Poston G, Ychou M, Rougier P; European Colorectal Metastases Treatment Group. Towards a pan-European consensus on the treatment of patients with colorectal liver metastases. Eur J Cancer. 2006 Sep;42(14):2212-21. doi: 10.1016/j.ejca.2006.04.012. Epub 2006 Aug 10. PMID 16904315
- [Background] Kemeny N, Huang Y, Cohen AM, Shi W, Conti JA, Brennan MF, Bertino JR, Turnbull AD, Sullivan D, Stockman J, Blumgart LH, Fong Y. Hepatic arterial infusion of chemotherapy after resection of hepatic metastases from colorectal cancer. N Engl J Med. 1999 Dec 30;341(27):2039-48. doi: 10.1056/NEJM199912303412702. PMID 10615075
- [Background] Tomlinson JS, Jarnagin WR, DeMatteo RP, Fong Y, Kornprat P, Gonen M, Kemeny N, Brennan MF, Blumgart LH, D'Angelica M. Actual 10-year survival after resection of colorectal liver metastases defines cure. J Clin Oncol. 2007 Oct 10;25(29):4575-80. doi: 10.1200/JCO.2007.11.0833. PMID 17925551
- [Background] Li ZQ, Liu K, Duan JC, Li Z, Su CQ, Yang JH. Meta-analysis of simultaneous versus staged resection for synchronous colorectal liver metastases. Hepatol Res. 2013 Jan;43(1):72-83. doi: 10.1111/j.1872-034X.2012.01050.x. Epub 2012 Sep 13. PMID 22971038
- [Background] Wei M, He Y, Wang J, Chen N, Zhou Z, Wang Z. Laparoscopic versus open hepatectomy with or without synchronous colectomy for colorectal liver metastasis: a meta-analysis. PLoS One. 2014 Jan 29;9(1):e87461. doi: 10.1371/journal.pone.0087461. eCollection 2014. PMID 24489916
- [Background] Arezzo A, Passera R, Scozzari G, Verra M, Morino M. Laparoscopy for rectal cancer reduces short-term mortality and morbidity: results of a systematic review and meta-analysis. Surg Endosc. 2013 May;27(5):1485-502. doi: 10.1007/s00464-012-2649-x. Epub 2012 Nov 25. PMID 23183871